CLINICAL TRIAL: NCT02509884
Title: Comprehensive Diagnosis and Treatment of Alveolar Echinococcosis : A Single-center, Longterm Observational Study of 312 Patients in Germany
Brief Title: Long-term Results of Comprehensive AE Management
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Beate Grüner, Beate Grüner, MD, University of Ulm
Other Study IDs: 166/13
Record Dates: First submitted 2015-07-12; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Alveolar Echinococcosis
Keywords: Alveolar Echinococcosis (AE); Echinococcus multilocularis; antiparasitic treatment; surgery; classification; staging; prospective cohort study
MeSH Terms: conditions — Alveolar echinococcosis; Echinococcosis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comprehensive diagnosis and treatment of Alveolar Echinococcosis : A single-center, long-term observational study of 312 Patients in Germany. Human alveolar echinococcosis (AE) is the most Iethal human helminthic infection and is one of the 17 neglected tropical diseases prioritized by the World Health Organization (WHO). Its incidence is low in endemic regions of Central and Western Europe (0.03-0.05/100,000), but morbidity and treatment costs are high. In this observational study, the investigators assessed the severity of the disease using the PNM staging system and report on the long-term results of specific AE therapy in an interdisciplinary team of clinicians.

DETAILED DESCRIPTION:
All patients with Alveolar Echinococcosis (AE) seen at the specialized treatment unit in Ulm between January 1992 and December 2011 were included in the database. Follow up ended on 31.12.2012. Cases were defined to the likelihood of diagnosis as a "possible", "probable" or "confirmed" case . Diagnosis of AE was based on clinical presentation, epidemiological history, pathognomonic imaging findings, specific laboratory results, such as immunodiagnosis or histopathological findings in resected/ biopsied specimens, and/or detection of nucleic acid sequences in such specimens. The location of the larval lesions and its spread at diagnosis was documented using the PNM classification. Treatment with benzimidazoles was followed the WHO-IWGE recommendations. Treatment efficacy was monitored by US examination and FDG-PET scan or MRI. To categorize each case at each visit the terms "cured", "stable" or "progressive" were used. Patients' data was assessed at each visit; missing information was obtained from hospital records or the family doctor. Names were anonymized and data was stored in a Microsoft Excel database. Statistics were done with SAS version 9.3.

The data were stratified into series A containing diagnoses until December 1999 and series B from January 2000 onwards. This separation was chosen as patient admissions to the clinic rose almost 3-fold in 2000 when notification of AE became mandatory in Germany. It can be assumed that series B better represents AE patient characteristics, disease manifestation and comprehensive management; series A includes case histories with favorable prognoses at the time of diagnosis while optimal treatment for AE was still unavailable.

Outcome parameters for this study population were: overall survival after diagnosis, relapse after surgery or progression of remaining liver lesions in size or new lesions in other organs, and time to relapse or progress. Survival was estimated by the Kaplan Meier method.

Parameters with an assumed influence on the time until relapse or progress of the parasitic lesions entered Kaplan Meier survival analysis and Cox proportional hazard regression model analysis, respectively, and hazard ratios (HR) with corresponding 95% confidence intervals (CI) were calculated. Logistic regression was used to identify factors which may predict a successful treatment interruption using the odds ratio (OR) as an appropriate outcome parameter.

ELIGIBILITY:
Inclusion Criteria:

* All patients with AE seen at the specialized treatment unit in Ulm between January 1992 and December 2011.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with AE seen at the specialized treatment unit in Ulm between January 1992 and December 2011 were included in the database. Follow-up ended on 31.12.2012. Cases were defined according to the likelihood of diagnosis as a "possible", "probable", or "confirmed case"
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 1992-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall survival after diagnosis, | inclusion January 1992-December 2011; end of follow-up December 2012 .Inclusion January 1992-December 1999 (series A).Inclusion January 2000- December 2011 (series B)
  Survival was estimated by the Kaplan Meier method.
Relapse after surgery or progression of remaining liver lesions in size or new lesions in other organs | inclusion January 1992-December 2011; end of follow-up December 2012.Inclusion January 1992-December 1999 (series A).Inclusion January 2000- December 2011 (series B)
  Parameters with an assumed influence on the time until relapse or progress of the parasitic lesions entered Kaplan Meier survival analysis and Cox proportional hazard regression model analysis, respectively, and hazard ratios (HR) with corresponding 95% confidence intervals (CI) were calculated.
Time to relapse or progress | inclusion January 1992-December 2011; end of follow-up December 2012.Inclusion January 1992-December 1999 (series A).Inclusion January 2000- December 2011 (series B)

SECONDARY OUTCOMES:
Symptoms and comorbidities | inclusion January 1992-December 2011; end of follow-up December 2012. Inclusion January 1992-December 1999 (series A).Inclusion January 2000- December 2011 (series B)
  Specific and unspecific symptoms were less frequent in case series B (44.6%) than in series A (61.1%; Table 4). 90 out of 204 (44.1 %) patients in B did not report any symptoms. Jaundice was more frequent in series A (17.6% vs. 7.8%). The occurrence of any kind of symptoms was closely associated with the disease stage: rates of patients with symptoms increased from 24.2% (stage I), to 32.6% (stage II), 50.8% (stage IIIa), 54.4% (stage IIIb) and 68.0% at stage IV. More cases in series A (56.7%) had no concomitant health problems when first diagnosed with AE. Notably, 18 cases of series B and 1 case of series A suffered from chronic inflammatory or immunologic syndromes including rheumatic disorders. 22 cases (7.1%) suffered from malignant diseases prior to AE diagnosis
Medical treatment and side effects | inclusion January 1992-December 2011; end of follow-up December 2012Inclusion January 1992-December 1999 (series A).Inclusion January 2000- December 2011 (series B)
  Side effects of medical therapy were monitored throughout follow-up, notably more closely during the first six months after start of ABZ. In cases of toxicity to the drug, postprandial ABZ sulfoxide plasma levels were used for guidance, and drug dose was reduced accordingly. For re-exposure ABZ was given at a lower dosage which was slowly raised over a period of one month. Patients with continuing toxicity were switched to MBZ. If toxicity remained, patients had prolonged medication pauses. Phases of non-adherence to the therapy regimen were noted if their duration was >3 months. Such phases due to drug intolerance, misunderstandings or non-compliance of the patients, were defined as "pauses".
Treatment interruption ant potential cure | inclusion January 1992-December 2011; end of follow-up December 2012.Inclusion January 1992-December 1999 (series A).Inclusion January 2000- December 2011 (series B)
  Treatment efficacy was monitored by US examination and, every 24 months, by alternating FDG-PET/CT scans and MRI.Structured treatment interruption was a goal for patients with an PanyN0M0 status at diagnosis, either after ascertained R0 resection and a two-year BMZ prophylaxis, as well as for patients with non-resectable lesions under the following assumptions 1) marked regression/absence of lesion(s) by imaging, 2) vanished enrichment of FDG around the AE lesion(s) assessed by FDG-PET/CT scan, 3) continuous BMZ medication for at least 2 years, 4) no extrahepatic involvement, 5) absence of any clinical symptoms or signs of illness, 6) marked changes in serology. Such medication-free phases were noted as "interruptions".
Surgical and interventional treatment | inclusion January 1992-December 2011; end of follow-up December 2012.Inclusion January 1992-December 1999 (series A).Inclusion January 2000- December 2011 (series B)
  After liver resections, surgical specimen was reviewed by the pathologist and graded as R0, R1, or R2 resections. Patients with R0 resections received ABZ for at least two years as "secondary prophylaxis" as recommended by WHO-IWGE (Anonymous 1996, Brunetti et al 2010). Drug treatment was indefinitely prescribed to patients after incomplete or palliative resections (R1 or R2), to all patients with extrahepatic lesions, and all cases with inoperable liver lesions. Some cases received BMZ days or weeks prior to surgery. Time on drug was noted as well as time on inappropriate dosage or pauses.

CONTACTS AND LOCATIONS:
Overall Officials: Beate Grüner, MD, Study Chair — University of Ulm

REFERENCES:
- [Background] Kern P, Wen H, Sato N, Vuitton DA, Gruener B, Shao Y, Delabrousse E, Kratzer W, Bresson-Hadni S. WHO classification of alveolar echinococcosis: principles and application. Parasitol Int. 2006;55 Suppl:S283-7. doi: 10.1016/j.parint.2005.11.041. Epub 2005 Dec 15. PMID 16343985
- [Background] Brunetti E, Kern P, Vuitton DA; Writing Panel for the WHO-IWGE. Expert consensus for the diagnosis and treatment of cystic and alveolar echinococcosis in humans. Acta Trop. 2010 Apr;114(1):1-16. doi: 10.1016/j.actatropica.2009.11.001. Epub 2009 Nov 30. PMID 19931502